CLINICAL TRIAL: NCT06769763
Title: Arabic Mobile Application for Multiple Sclerosis (MS) Patients and Its Effect on Their Quality of Life and Self-care Practices
Brief Title: MHealth Effect on Multiple Sclerosis Patients' Quality of Life and Self-care Practices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Emeash, Assistant lecturer of Public Health and Community Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MD-204-2024
Record Dates: First submitted 2025-01-09; First posted 2025-01-10 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Quality of life; Self-care; mHealth; Arabic Application
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- App users (Active Comparator): This arm is the interventional group who will use the application for 3 months
  Interventions: Other: My Journey with MS application
- Control arm (No Intervention): This arm will not use the application during the period of follow-up.

INTERVENTIONS:
Other: My Journey with MS application — This is an Arabic application for MS patients that provides them with information about self-care like nutrition, exercise, mental health, and self-management, in addition to other features like symptom tracking and medication reminders.
  Arms: App users

SUMMARY:
The goal of this clinical trial is to learn if an Arabic mobile application for multiple sclerosis patients will improve self-care practice and the quality of life of patients or not. The main question it aims to answer is:

Does the Arabic mobile application for MS patients will improve their self-care and quality of life?

Participants will:

Use the developed application or usual care without using the application for 3 months Be followed up during the 12 week period and asked to follow the instructions in the application

DETAILED DESCRIPTION:
This study aims to build and test a culturally appropriate mobile application in Arabic for MS (multiple sclerosis) patients in Egypt. It will focus on self-care practices and quality of life enhancement via educational material provision, symptom tracking as well as medication adherence reminders among other possible functions depending on user preferences. The study shall evaluate how effective the developed app is in promoting self-care practices and improving the quality of life for MS patients compared to a control group who do not use the app.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed clinically with multiple sclerosis.
* From 18 to 50 years old (adult).
* With smartphones.
* Willing to participate in the study and use the mobile application.

Exclusion Criteria:

* Patients who are bedridden or in a wheelchair
* Illiterate patients.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
The effect of mHealth on the self-care practices of multiple sclerosis patients | From enrollment to the end of follow-up at 12 weeks
  The effect of mHealth on the self-care practices of multiple sclerosis patients will be assessed using the self-care for chronic disease inventory questionnaire. The score ranges from 0 to 100, the higher the score the better the self-care practices.
The effect of mHealth on the quality of life of multiple sclerosis patients | From enrollment to the end of follow-up at 12 weeks
  The effect of mHealth on the quality of life (QoL) of multiple sclerosis patients will be assessed using the multiple sclerosis international quality of life (Musiqol) questionnaire. The score will be transformed into a range from 0 to 100; the higher the score, the better the QoL practices.

SECONDARY OUTCOMES:
The usability of the developed application | After 12 weeks of enrollment
  The usability of the developed application will be assessed using the app usability questionnaire. The patients will choose a number between 1 to 7 (Likert scale), as 1 strongly disagree, 2 disagree, 3 somewhat disagree 4 neutral, 5 somewhat agree, 6 agree, and 7 strongly agree. Then the total average of all scored items for each participant will be calculated; the higher the average, the better the app's usability

CONTACTS AND LOCATIONS:
Overall Officials: Nargis Albert Labib, Study Chair — Professor of public Health and Community Medicine, Faculty of Medicine, Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
The information may not be shared if it violates the data's confidentiality, and can't be ensured that it will not be used for purposes not present in the consent form.